CLINICAL TRIAL: NCT03132649
Title: Impact of Three-dimensional Visualization on Operation Strategy and Complications for Hilar Cholangiocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201701
Record Dates: First submitted 2017-04-09; First posted 2017-04-28 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-02

CONDITIONS: Hilar Cholangiocarcinoma
Keywords: Three dimensional visualization; Operation strategy
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The biospecimen will be comformed by histopathological examination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the multi-centre study is to evaluate correctly the impact of three-dimensional visualization on operation strategy and complications for hilar cholangiocarcinoma.

DETAILED DESCRIPTION:
Because of the complexity of hilar cholangiocarcinoma,the limitations of 2D images of CT/MRI and the uncertainty of surgeons'experience, it is difficult for the surgeons to diagnosis and assess the operation strategy accurately based on traditional 2D imaging(CT/MRI).The aim of the multi-centre study is to evaluate correctly the impact of three-dimensional visualization on operation strategy and complications for hilar cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years≤ Age ≤70 years
2. Complying with the diagnosis criteria of hilar cholangiocarcinoma.
3. Without intrahepatic or extrahepatic extensive cancer metastasis.
4. Preoperative serum bilirubin ≤51.3 umol/L or preoperative serum bilirubin < 200 umol/L after the drainage by PTCD(percutaneous transhepaticcholangial drainage)/ENBD(endoscopic nasobiliary drainage).
5. The patients are volunteered for the study.

Exclusion Criteria:

1. Patients with mental illness.
2. Patients can't tolerate the operation owe to a variety of basic diseases (such as severe cardiopulmonary insufficiency, renal insufficiency, cachexia and blood system diseases, etc.)
3. The patients refused to take part in the study.
4. There are other co-existed malignant tumors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with hilar cholangiocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Impact on operation strategy of three-dimensional visualization technique | 2 year
  Firstly, the operation strategies based on original CT or MRI image data will be made by the team, Secondly, the operation strategies based on three dimensional reconstruction models will be made by the team, then, actually surgical strategies will be recorded. The change of operation strategy will be assessed by comparing the strategy of the 2D model and 3D model. The change rate of operation strategy will be recorded and presented as percentage.
Impact on complications of three-dimensional visualization technique | 2 year
  The complications are refer to the classification of Clavien-Dindo, including postoperative bleeding, biliary fistula, ascites, postoperative liver failure, renal dysfunction, pleural effusion, abdominal cavity infection, abdominal abscess, incision infection, the occurrence cases of each complications (number) will be recorded.

SECONDARY OUTCOMES:
Blood routine examination (the 1th, 3 th, 5th, 7th) | 2 year
  Hemoglobin(g/L), Platelet(109/L), and neutrophilic granulocyte percentage (%)
Urine routines (the 1th, 3 th,5th, 7th) | 2 year
  Urine specific gravity, urine protein(mg/dl), urine sugar(mmol/L), leukocytes in urine(number/ul), urine erythrocyte(number/ul)
Stool Routine (the 1th, 3 th,5th, 7th) | 2 year
  Defecate occult blood test, Microorganisms (mold, parasites, etc.)
Blood biochemistry (the 1th, 3 th,5th, 7th) | 2 year
  Serum albumin(g/L), serum pre-albumin(g/L), serum globulin(g/L), total bilirubin(µmol/L), direct bilirubin(µmol/L),serum glutamic-oxaloacetic transaminase (AST, IU/L), serum glutamic pyruvic transaminase (ALT, IU/L), alkaline phosphatase (ALP, IU/L), gamma glutamyl transpeptidase（r-GGT, IU/L） ,Serum creatinine(µmol/L), Urea(mmol/L), Blood sugar(mmol/L)
Tumor marker | 2 year
  Alpha fetoprotein(AFP, ng/L), Carbohydrate antigen-199(CA-199, ku/L), Carbohydrate antigen-125(CA-125, ku/L), Carcinoembryonic antigen (CEA, ng/L), Carbohydrate antigen-153(CA-153, ku/L)
The blood coagulation function (the 1th, 3th, 5th, 7th) | 2 year
  prothrombin time (PT, s), partial thromboplastin time (APTT), international normalized ratio (INR), plasma prothrombin activity (PTA, %), fibrinogen (FIB, g/L), d-dimer(mg/L)
Inflammatory biomarkers | 2 year
  C-reactive protein, procalcitonin
Preoperative viral loading | 2 year
  HBV(hepatitis B virus)- DNA、HCV(hepatitis C virus)- RNA
Postoperative results of paraffin wax and immunohistochemical index | 2 year
  CK7、CK18、CK19、Hepatocyte、CD34（vascular）、S-100（nerve）、D2-40（lymphatic）、AFP、Ki67
Postoperative pathologic examination | 2 year
  The stage of TNM, The condition of resection (R0/R1/R2), the condition of liver cirrhosis, the pathological type of the tumor (Nipple type/nodule type/infiltration type)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No